CLINICAL TRIAL: NCT06025760
Title: Evaluation of Diaphragmatic Function and Quadriceps Muscle Thickness Using Ultrasonography in Critically Ill Mechanically Ventilated Patients Receiving High Protein Nutrition
Brief Title: Evaluation of Diaphragmatic Function and Quadriceps Muscle Thickness in Patients Receiving High Protein Nutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Naglaa Fathy Abdelhaleem Abdelhaleem, Lecturer of anesthesia and ICU, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB#9659
Record Dates: First submitted 2022-12-06; First posted 2023-09-06 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: ICU Acquired Weakness

STUDY DESIGN:
Intervention Model Description: Critically ill mechanically ventilated patients will receive protein of 2 gm/kg/day in the interventional group. Critically ill mechanically ventilated patients will receive protein of 1.2 gm/kg/day in the control group.
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Active Comparator): Mechanically ventilated patients will receive a nutritional caloric intake of 25-30 kcal/kg/day with a high protein dose of 2 gm protein /kg/day within 24 hours of ICU admission.
  Interventions: Other: patients who will receive 2 gm protein/kg/day will be evaluated by ultrasound for diaphragmatic function and quadriceps muscle thickness
- Control group (Placebo Comparator): patients will receive a nutritional caloric intake of 25-30 kcal/kg/day with a standard protein dose of 1.2 gm protein /kg/day within 24 hours of ICU admission.
  Interventions: Other: patients who will receive 2 gm protein/kg/day will be evaluated by ultrasound for diaphragmatic function and quadriceps muscle thickness

INTERVENTIONS:
Other: patients who will receive 2 gm protein/kg/day will be evaluated by ultrasound for diaphragmatic function and quadriceps muscle thickness — All patients after ICU admission will be started enteral nutrition through a nasogastric tube within 24-48 hours. The target caloric intake is 25-30 kcal/kg/day. patients in the interventional group will receive 2 gm protein/kg/day, while patients in the control group will receive 1.2 gm protein/kg/day. Quadriceps thickness and Diaphragm thickening fraction will be assessed by ultrasound from the time of admission on days 0, 3, 5, and 7 then weekly till the fourth week.
  Other Names: patients who will receive 1.2 gm protein/kg/day will be evaluated by ultrasound for diaphragmatic function and quadriceps muscle thickness in

SUMMARY:
Different Protein Doses' Effect on Diaphragmatic Function and Quadriceps Thickness

DETAILED DESCRIPTION:
Nutrition therapy is no longer a support method for critically ill patients but is considered an important treatment measure. Increasing the protein and energy available to patients in the intensive care unit (ICU) reduces infection and complications, increases ventilator-free days, increases long-term physical recovery, and lowers patient mortality Among critically ill patients, protein is the most important macronutrient because it promotes healing, improves immune function, and helps patients maintain their lean body mass. Growing evidence has shown that adequate protein intake may be more important than caloric intake in the body. In addition, reaching at least 80% of the prescribed protein intake rather than energy intake is related to improved survival rates in ICU patients.

Muscular atrophy is a common feature in patients with intensive care unit-acquired weakness (ICU-AW), and it can start in the early stages of critical illness (within hours of onset of the disease). Its development has been related to the acute inflammatory process and immobilization. Factors such as age, medications, comorbidities, nutrition, and nervous, and muscular damage before critical illness can contribute to the extent of atrophy and the muscular and functional recovery capacity.

It was believed that perhaps the respiratory muscles in humans were spared any loss of muscle protein during starvation because of their constant activity. In a necropsy study designed to assess the diaphragm in health and disease, it was found that alterations in body weight and muscularity profoundly affect the diaphragm muscle mass.

Mechanical ventilation (MV) is the most important life-sustaining measure for critically ill patients, Even if the MV is maintained for a short time, diaphragm fatigue may also occur owing to atrophy or decreased contractile function, which is known as ventilator-induced diaphragm dysfunction (VIDD). Pathophysiological changes of VIDD include muscle atrophy, structural damage, and fiber-type transformation and remodeling.VIDD is the main factor contributing to difficult weaning from long-term MV in critically ill patients. Prolonging the time of MV is associated with an increased risk of complications, long-term dysfunction, and death.

Muscles of the lower limb are more prone to early atrophy as they are weight-bearing compared to the muscles of the upper limb as shown in previous studies. The authors showed that the size of the flexor compartment of the elbow did not show any change in the first 10 days of admission, whereas the size of the anterior compartment muscles of the lower limb showed a greater decrease in thickness within the first 5 days. Thus, these muscles make a good choice for muscle mass assessment.

Point-of-care ultrasound (POCUS) is rapid, accurate, repeatable, nonexpensive, noninvasive, and without the risk of radiation. It can visualize a large muscle area and deeper-located muscles. It can be used in both stable and unstable patients. Performing repeated ultrasound examinations in critical patients is essential and improves the overall sensitivity of the examination, which has become a standard of care in critical care.

One of the unsolved problems for a reliable definition of protein goals is the optimal intake timing to reach predefined therapeutic goals. European Society for Clinical Nutrition and Metabolism (ESPEN) 2009 recommended protein dose to be 1.2 - 1.5 gm /kg/day, while recent ESPEN 2019 guidelines recommend a dose of 1.3 gm/kg/day. On the other hand, the American Society for Parenteral and Enteral Nutrition (ASPEN) 2016 and ASPEN 2022 recommend a dose of 1.2- 2 gm/kg/day.

Generally, it is well known that patients in the acute phase (ebb phase) of the stress response are less capable of utilizing nutrients, thereby implying that early high-dose protein administration might not be beneficial. In the later phase (flow phase) of metabolic stress, insulin sensitivity gradually improves, and the human body's capability to metabolize exogenous substrates increases accordingly.

ELIGIBILITY:
Inclusion Criteria:

* • Acceptance of the first-degree relatives.

  * Critically ill patients: patients with a life-threatening condition that requires pharmacological and/or mechanical support of vital organ functions without which death would be imminent.
  * Patients anticipated to be mechanically ventilated for ≥ 48 hours
  * Patients who expected ICU stay ≥ 4 weeks
  * Patients aged between 18 - 60 years of both sexes.
  * Patient nutrition risk screening (NRS 2002) score ≥ 3
  * Patient BMI less than 35
  * No contraindication to early enteral nutrition.

Exclusion Criteria:

* • Patient with Trauma to both lower extremities, diaphragm disease (trauma, immobilization….), myopathy, and moderate to severe hepatic insufficiency.

  * Patient receiving steroids.
  * Patient on renal replacement therapy.
  * Prior MV before admission.
  * Pregnant.
  * Patient with neuromuscular disease, spinal cord injury, thoracic deformity, and respiratory restriction.
  * Patients require muscle paralysis on MV.
  * Patients require high dose inotrope or vasopressor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
To assess the effect of different protein doses (1.2 gm/kg per day versus 2 gm/kg per day ) on diaphragmatic muscle function in mechanically ventilated patients in ICU for 4 weeks. | from time of ICU admission on day 0,then on days 3, 5, 7, then weekly till the fourth week.
  assessment of the effect of different protein doses per day on diaphragmatic muscle function in mechanically ventilated patients using ultrasound, the following data will be assessed:
  1. Diaphragm thickness (mm) on days (0, 3, 5, and 7 from ICU admission then weekly till the fourth week ).
  2. Diaphragm thickening fraction on the day (0, 3, 5, 7 then weekly till the fourth week )
  3. Diaphragm excursion during the weaning trial during spontaneous breathing trial (SBT).

SECONDARY OUTCOMES:
To assess the effect of different protein doses (1.2 gm/kg per day versus 2 gm/kg per day ) on Quadriceps muscle thickness(mm) in mechanically ventilated patients in ICU for 4 weeks. | from time of ICU admission on day 0, then on days 3, 5, 7, then weekly till the fourth week
  Assessment of the effect of different protein doses per day on quadriceps muscle layer thickness (mm) in mechanically ventilated patients in ICU using ultrasound, the following data will be assessed :
  Quadriceps muscle layer thickness on the day (0, 3, 5, 7, from ICU admission then weekly till the fourth week )

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Abdelrazik, professor, Study Chair — Professor of anesthesia, intensive care and pain managment; Neven Gamil, professor, Study Chair — Professor of anesthesia, intensive care and pain managment; Naglaa Abdelhaleem, Lecturer, Study Chair — lecturer of anesthesia, intensive care and pain managment; Ayman Amer, professor, Study Chair — Professor of diagnostic radiology

IPD SHARING:
Plan to Share IPD: No
Not decided yet